CLINICAL TRIAL: NCT05137704
Title: Healthcare Resources Utilization and Associated Costs of Adult ADHD in England
Brief Title: A Study on the Use of Healthcare Resources and Costs of Attention Deficit Hyperactivity Disorder (ADHD) in Adults in England
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-489-4005
Record Dates: First submitted 2021-11-25; First posted 2021-11-30 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant With ADHD: The record available for ADHD participants in primary care-based electronic medical records in the CPRD database linked to secondary care based episodic claims data available in HES database will be assessed.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a non-interventional study.

SUMMARY:
The main aim of the study is to learn about the demographic and clinical characteristics, healthcare resources utilization (HCRU) and costs associated with before and after ADHD diagnosis in England. No study medicines will be provided to participants in this study. The record available in Clinical Practice Research Datalink (CPRD) database and Hospital Episode Statistics (HES) database for ADHD participants will be assessed.

ELIGIBILITY:
Inclusion Criteria

1. Age greater than or equal to (>=) 18 years at the beginning of the patient observation period (that is 18-months prior to the adult ADHD diagnosis to ensure they would have been seen in adult health care services).
2. First record of an adult ADHD diagnosis between 01st January 2016 and 30th June 2018.
3. Data availability in the database at least during the 18-months before and after the index date.

Exclusion Criteria

A participant will be excluded from the study if their CPRD linked to HES electronic medical record data includes:

1. Incomplete information for key demographics (that is, missing age or sex).
2. Clinical history of a diagnosis of ADHD during childhood or adolescence.
3. Prescription of a licensed adult ADHD medication (that is, methylphenidate, lisdexamfetamine, dexamfetamine, atomoxetine) during the pre-index period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant diagnosed with ADHD recorded between 01 January 2016 and 30 June 2018.
Sampling Method: Non-Probability Sample
Enrollment: 2236 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Number of General Practitioner (GP) Appointments | Up to approximately 36 months
  Number of GP appointments will be reported.
Number of Referrals to Psychiatrist | Up to approximately 36 months
  Number of referrals to psychiatrist will be reported.
Number of Referrals by Specialist | Up to approximately 36 months
  Number of referrals by specialist will be reported.
Number of Outpatient Visits by Specialist | Up to approximately 36 months
  Number of outpatient visits by specialist will be reported.
Number of Investigations Undergone | Up to approximately 36 months
  Number and type of investigations undergone will be reported.
Number of Accident and Emergency Visits | Up to approximately 36 months
  Number of accident and emergency visits will be reported.
Number of Reasons for Admission | Up to approximately 36 months
  Number of reasons for admission will be reported.
Number of Inpatient Hospitalizations | Up to approximately 36 months
  Number of inpatient hospitalizations will be reported.
Length of Stay in Hospital | Up to approximately 36 months
  Length of stay in hospital will be reported.
Total Healthcare Costs | Up to approximately 36 months
  Health care cost includes prescription costs, primary health care consultations, investigations, hospital admissions, and outpatient appointments.
Number of Participants Prescribed With Pharmacological Treatments | Up to approximately 36 months
  Number of participants prescribed with pharmacological treatment will be reported.
Number of Participants Received Non-Pharmacological Treatments | Up to approximately 36 months
  The number of participants who received non-pharmacological treatments will be reported.
Number of Participants Received Non-Pharmacological Therapy | Up to approximately 36 months
  The non-pharmacological therapy will be cognitive behavioural therapy. Number of participants who received non-pharmacological therapy will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- IQVIA Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61a6927bf571d4002a64b43a